CLINICAL TRIAL: NCT00196807
Title: Prostate Cancer Screening: Fostering Informed Decisions
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Kathryn L. Taylor, PhD, Principal Investigator, Georgetown University Medical Center
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: R01CA098967 (NIH); R01CA098967 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2010-01

CONDITIONS: Prostate Cancer
Keywords: prostate cancer screening; medical decision making; informed decision making; patient education; male
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Information plus DA at home (Experimental)
  Interventions: Behavioral: patient decision aid (print-based)
- UC Information at home (Active Comparator)
  Interventions: Behavioral: patient decision aid (print-based)
- Information plus decision aid at clinic (Experimental)
  Interventions: Behavioral: patient decision aid (print-based)
- UC Information at clinic (Active Comparator)
  Interventions: Behavioral: patient decision aid (print-based)

INTERVENTIONS:
Behavioral: patient decision aid (print-based) — To evaluate the impact of the decision aid intervention (information plus decision aid (IDA) vs. usual care (UC)), and timing of intervention delivery (at Home (pre-screening) vs. in the Clinic (screening day)) on key patient outcome variables of PCa knowledge and decisional satisfaction.
  Other Names: Information plus Decision Aid at home; Information plus Decision Aid at clinic; Usual Care at home; Usual Care at clinic

SUMMARY:
The primary goal of this study is to develop and evaluate a print-based method of patient education with a decision tool that is designed to provide detailed information about prostate cancer and to clarify patient preferences and values, ultimately assisting men in making an informed screening decision.

DETAILED DESCRIPTION:
In spite of the significant disease burden presented by PCa, the utility of screening asymptomatic men remains controversial, as it has not yet been demonstrated by a randomized trial that early diagnosis and treatment of PCa reduces disease-related mortality. The primary goal of the proposed study is neither to encourage nor discourage PCa screening, but to evaluate a method of patient education that is designed to provide detailed screening and treatment-related information and to clarify patient preferences and values, ultimately assisting men in making an informed screening decision. The target population for this educational intervention will be men who have registered to undergo PCa screening within a free, mass screening program. Although at first this may appear to be an atypical group to target for an educational intervention, we present information suggesting that this population represents a large and uniformed group for whom effective and inexpensive methods of education are of critical importance. We will test the impact of providing men with detailed information and a decision aid vs. usual care information and the impact of the timing of administration of information (a week or more prior to the screening vs. usual care, which is on the day of screening). Participants will include men who register for the annual PCa mass screening programs held at Georgetown University and at Howard University during the 2004 and 2005 screening programs. Following enrollment and the baseline interview, participants will be randomly assigned to one of four groups: 1) Information plus Decision Aid received prior to the scheduled screening date (IDA-home); 2) Information plus Decision Aid received on the day of screening (IDA-clinic); 3) Usual Care information received prior to the scheduled screening date (UC-home); or 4) Usual Care information received on the day of the screening (UC-clinic). Follow-up assessments will be conducted post-screening, post receipt of screening results, and one-year post-intervention, to measure knowledge, decisional conflict, decisional satisfaction, and the actual screening decision. We will utilize a 2 (IDA/UC) X 2 (Home/Clinic) X 2 (AA/white) repeated measures analysis of covariance to assess for group differences on these outcomes. If found to be effective, the long-term goal of this research program is to disseminate this informational decision aid for use in mass screening programs.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria are: 1) 40-70 years old, 2) English-speaking, and 3) ability to provide meaningful consent.

Exclusion Criteria:

* The exclusion criteria are: 1) a history of cancer (with the exception of basal cell carcinoma), and 2) a history of prostate disease that has required treatment (e.g., benign prostatic hypertrophy).

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 543 (Actual)
Dates: Start 2004-08; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Patient knowledge and decisional satisfaction measured at one month following the intervention. | one-month and one-year follow-up assesments

SECONDARY OUTCOMES:
Decisional conflict measured at one month and the screening decision measured at one year post intervention. | one-month and one-year follow-up assesments

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn L. Taylor, Ph.D., Principal Investigator — Georgetown University
Locations (2):
- United States (2):
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Howard University Hospital, Washington D.C., District of Columbia

REFERENCES:
- [Background] Taylor KL, Africano NL, Schwartz M, Cullen J, Ahaghotu C. Prostate cancer screening at National Cancer Institute comprehensive and clinical cancer centers. J Natl Cancer Inst. 2004 Mar 3;96(5):414-5. doi: 10.1093/jnci/djh073. No abstract available. PMID 14996868
- [Result] Red SN, Kassan EC, Williams RM, Penek S, Lynch J, Ahaghotu C, Taylor KL. Underuse of colorectal cancer screening among men screened for prostate cancer: a teachable moment? Cancer. 2010 Oct 15;116(20):4703-10. doi: 10.1002/cncr.25229. PMID 20578178
- [Derived] Taylor KL, Williams RM, Davis K, Luta G, Penek S, Barry S, Kelly S, Tomko C, Schwartz M, Krist AH, Woolf SH, Fishman MB, Cole C, Miller E. Decision making in prostate cancer screening using decision aids vs usual care: a randomized clinical trial. JAMA Intern Med. 2013 Oct 14;173(18):1704-12. doi: 10.1001/jamainternmed.2013.9253. PMID 23896732